CLINICAL TRIAL: NCT04979325
Title: A Study on the Application Status of Extracorporeal Membrane Oxygenation (ECMO) in Zhejiang Province
Brief Title: Cross-sectional Survey of Zhejiang ECMO Application
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Zhejiang Provincial People's Hospital (Other); Zhejiang Hospital (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); First People's Hospital of Hangzhou (Other); The Affiliated Hospital of Hangzhou Normal University (Other); The Third People's Hospital of Hangzhou (Other); Red Cross Hospital, Hangzhou, China (Other); Hangzhou Children's Hospital (Unknown); The First Hospital of Fuyang District, Hangzhou (Unknown); The First Hospital of Xiaoshan District, Hangzhou (Unknown); The First Hospital of Linping District, Hangzhou (Unknown); The First Hospital of Lin'an District, Hangzhou (Unknown); The First Hospital of Tonglu County, Hangzhou (Unknown); The First Hospital of Jiande County, Hangzhou (Unknown); The First Hospital of Chun'an County, Hangzhou (Unknown); Affiliated Cixi Hospital of Wenzhou Medical University (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Ningbo First People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: I2021001538
Record Dates: First submitted 2021-06-07; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-06

CONDITIONS: Extracorporeal Membrane Oxygenation; Cardiopulmonary Resuscitation; Epidemiology
Keywords: Extracorporeal membrane oxygenation; Epidemiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Extracorporeal lung oxygenation (ECMO) was first used in neonates in the 1970s and is now widely used to treat adult patients with intractable shock and respiratory failure who have failed various types of conventional life support. According to the Extracorporeal Life Support Organization (ELSO), a total of 61,193 adult patients worldwide received ECMO in 2019. According to the Extracorporeal Life Support Organization (ELSO), a total of 61,193 adult patients were treated with ECMO worldwide in 2019, including 25,631 VV-ECOM, 12,836 VA, and 5086 ECPR. The number of ECMO cases and hospitals in Zhejiang province are increasing year by year, and they play an irreplaceable role in various critical care resuscitation, especially in response to public emergencies, but there is a lack of precise data on the current status of ECMO implementation. This study aims to investigate the implementation of ECMO, problems and needs of hospitals at all levels in Zhejiang Province, and provide reference for further improving the capacity and quality of ECMO application in the province.

DETAILED DESCRIPTION:
This is a multicenter cross-sectional survey study ,was conducted jointly by the Zhejiang Emergency Medicine Quality Control Center, the Zhejiang Medical Emergency Medicine Branch and the Zhejiang Physicians Association Emergency Physicians Branch. The survey covers the general situation and ECMO implementation in general public hospitals at the county and district level in Zhejiang Province, including people's hospitals, Chinese medicine hospitals and above.

ELIGIBILITY:
Inclusion Criteria:

* All general hospitals at the first people's hospital and above at the county and district level in Zhejiang Province

Exclusion Criteria:

* Hospitals that explicitly do not wish to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All general hospitals at the first people's hospital and above at the county and district level in Zhejiang Province
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Contains the general description of the hospital | 1 year
  including hospital level, nature, number of approved beds, total number of outpatient and emergency departments in 2019, number of discharges, and number of operations
ECMO configuration | 1 year
  ECMO equipment manufacturers, models, number of ECMOs, belonging departments, and those who are proficient in ECMO Health care team
ECMO development status | 1 year
  first case development time, independent hospital development time, number, type and number of weaning machines carried out in 2019, operating costs, etc

SECONDARY OUTCOMES:
Zhejiang Hospital's Cognitive Status of ECMO Development | 1 year
  The surveyed unit's views on ECMO's role in hospitals, discipline development and the rescue of critically ill patients, the main difficulties encountered in carrying out ECMO, and the need for ECMO training and quality control

CONTACTS AND LOCATIONS:
Overall Officials: Bin Zhang, masters, Principal Investigator — Departmental staff
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine & Institute of Emergency Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No